CLINICAL TRIAL: NCT06039319
Title: Acute Effects of Maternal Exercise and the Growth Restricted Pregnancy
Status: Completed | Type: Observational
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 4967
Record Dates: First submitted 2023-07-11; First posted 2023-09-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2023-09

CONDITIONS: Fetal Growth Retardation; Fetal Growth Complications; Placental Insufficiency
MeSH Terms: conditions — Fetal Growth Retardation; Placental Insufficiency | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Appropriate Growth: Pregnant individuals with normal estimated fetal weight
  Interventions: Other: Physical activity
- Fetal Growth Restricted: Pregnant individuals with fetal growth restriction
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Physical activity — 30 minute bout of moderate intensity physical activity performed on a treadmill

SUMMARY:
Objectives / Specific Aims

* The purpose of this study is to investigate the acute effects of a single bout of moderate intensity maternal exercise on fetal well-being in a pregnancy affected by fetal growth restriction. Fetal well-being will be measured by biophysical profile (BPP), non-stress test (NST) and umbilical artery dopplers.
* The hypothesis is that a single bout of maternal exercise will not significantly alter fetal well-being or fetal status.

DETAILED DESCRIPTION:
Background and Significance

Regular exercise during pregnancy is beneficial in many ways, including decreased rates of diabetes or hypertensive disorders and decreased risks of preterm birth and cesarean deliveries. Many people use exercise to treat anxiety and depression as well as meet gestational weight gain recommendations. Regular exercise, defined as 150 minutes of moderate intensity exercise per week, is recommended in uncomplicated pregnancies. In some summary statements, fetal growth restriction (FGR) is noted as a relative or absolute contraindication to regular exercise. The American College of Obstetrics and Gynecology (ACOG), however, does not list FGR as a contraindication to maternal exercise. Currently, there are few high-quality studies about the effect of a recommended amount of maternal exercise on acute fetal status in pregnancies affected by FGR. The existing theories conflict. One theory is that maternal exercise will divert blood flow away from the uterus/fetus which could be deleterious in an already compromised pregnancy. The other theory is that exercise increases cardiac output and would therefore increase blood flow to the fetus. A previous study evaluated growth restricted fetuses after a single 5-minute bout of maternal exercise. This study population was heterogenous and used non-standardized measures of fetal assessment, making the results difficult to clinically interpret. In a previous study of healthy pregnancies, 30 minutes of moderate maternal exercise has been determined to have no effect on acute fetal status. The current study seeks to understand the acute fetal response to a single maternal exercise episode in pregnancies affected by FGR.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria - FGR population

  * Age 18-45
  * Intrauterine pregnancy with diagnosis of fetal growth restriction (FGR) as defined by total estimated fetal weight <10%ile for EGA or abdominal circumference <10%ile for EGA
  * Diagnosis of FGR at any point in gestation (preference given for inclusion of those diagnosed with FGR after 32w0d)
  * Gestational age between 28w0d and 36w6d at time of intervention (based on sure last menstrual period (LMP) confirmed by first or second trimester ultrasound or unsure LMP with first trimester ultrasound)
  * Compliant with standard prenatal care

Inclusion Criteria - Average for gestational age (AGA) population

* Age 18-45
* Intrauterine pregnancy with normal estimated fetal growth (EFW >10%ile and <90%ile)
* Gestational age between 28w0d and 36w6d at time of intervention with accurate dating (based on sure LMP confirmed by ultrasound prior to 22 weeks or unsure LMP with first trimester ultrasound)
* Compliant with standard prenatal care

Exclusion Criteria:

* Exclusion Criteria - FGR population

  * Known contraindication to completion of 30 minutes of moderate intensity exercise
  * Fetal umbilical artery with elevated S/D ratio or absent or reversed diastolic flow
  * BMI >40
  * Severe maternal anemia (Hb less than 8.0)
  * Placenta previa
  * 2nd or 3rd trimester vaginal bleeding
  * Preterm premature rupture of membranes
  * Cervical insufficiency
  * Multi-fetal gestation
  * Oligohydramnios
  * Hypertensive disorder requiring antihypertensive medication
  * Blood pressure >140/90 on the day of the study visit prior to exercise
  * Tobacco use
  * Opioid agonist therapy
  * Known fetal chromosomal anomaly, structural anomaly or infection
  * Inability or unwillingness of subject to give informed consent
  * Current psychiatric illness/social situation that would limit compliance with study requirements, as determined by the principle investigators

Exclusion Criteria - AGA population

* Known contraindication to completion of 30 minutes of moderate intensity exercise
* BMI >40
* Severe maternal anemia (Hb less than 8.0)
* Placenta previa
* 2nd or 3rd trimester vaginal bleeding
* Preterm premature rupture of membranes
* Cervical insufficiency
* Multi-fetal gestation
* Oligohydramnios
* Hypertensive disorder requiring antihypertensive medication
* Blood pressure >140/90 on the day of the study visit prior to exercise
* Tobacco use
* Opioid agonist therapy
* Known fetal chromosomal anomaly, structural anomaly or infection
* Inability or unwillingness of subject to give informed consent
* Current psychiatric illness/social situation that would limit compliance with study requirements, as determined by the principle investigators

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant individuals, between 28 weeks 0 days and 36 weeks 6 days gestational age with AGA or FGR.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in umbilical artery dopplers systolic/diastolic ratio from pre to post exercise | Pre to immediately post acute exercise
  Change in physiological assessment of umbilical artery dopplers systolic/diastolic ratio measured using ultrasound

SECONDARY OUTCOMES:
Change in uterine artery dopplers from pre to post exercise | Pre to immediately post acute exercise
  Change in physiological assessment of uterine artery dopplers measured using ultrasound
Change in fetal middle cerebral arterial (MCA) dopplers pulsatility index from pre to post exercise | Pre to immediately post acute exercise
  Change in physiological assessment of fetal middle cerebral arterial (MCA) dopplers pulsatility index measured using ultrasound
Biophysical Profile (BPP) pre exercise | Pre exercise (within 1 hour of the start of acute exercise bout)
  Physiological assessment of Biophysical Profile (BPP) pre exercise using ultrasound, which assesses and scores fetal wellbeing in the following areas: body movement, muscle tone, breathing movements, and amniotic fluid volume. Each component of the biophysical profile receives a score of 0-2, with a total potential score ranging from 0-8. A score of 0 reflects fetal a fetal emergency and/or ominous fetal status and a score of 8 is regarded as "reassuring" which means normal.
Time to complete Biophysical Profile (BPP) pre exercise | Pre exercise (within 1 hour of the start of acute exercise bout)
  Time to complete physiological assessment of Biophysical Profile (BPP) pre exercise.
Biophysical Profile (BPP) post exercise | Immediately post acute exercise
  Physiological assessment of Biophysical Profile (BPP) post exercise using ultrasound, which assesses and scores fetal wellbeing in the following areas: body movement, muscle tone, breathing movements, and amniotic fluid volume. Each component of the biophysical profile receives a score of 0-2, with a total potential score ranging from 0-8. A score of 0 reflects fetal a fetal emergency and/or ominous fetal status and a score of 8 is regarded as "reassuring" which means normal.
Time to complete Biophysical Profile (BPP) post exercise | Immediately post acute exercise
  Time to complete physiological assessment of Biophysical Profile (BPP).
Change in blood glucose from pre to immediately post acute exercise | Pre (within 1 hour of the start of acute exercise bout) to immediately post acute exercise
  Change in physiological assessment of capillary blood glucose measured using glucometer
Change in blood lactate from pre to immediately post acute exercise | Pre (within 1 hour of the start of acute exercise bout) to immediately post acute exercise
  Change in physiological assessment of capillary blood lactate using lactate analyzer
Change in maternal mood | Pre (within 1 hour of the start of acute exercise bout) to 20 minutes post exercise
  Change in maternal mood using the Brunel Mood Scale Questionnaire. The Brunel Mood Scale is a 32-item questionnaire of current mood descriptors, assessed via 5-point Likert scale questions ("not at all" 0 to "extremely" 4). Mood descriptors are arranged into 8 different subscales (anger, confusion, depression, fatigue, tension, vigor, happiness, calmness), which have a scoring range from 0-16. Higher scores correspond to greater presence of the subscale.
Change in maternal anxiety | Pre (within 1 hour of the start of acute exercise bout) to 20 minutes post exercise
  Change in maternal anxiety using the State Trait Anxiety Inventory (STAI) forms Y1 (20 items) and Y2 (20 items) which assess state and trait anxiety. Each STAI item is given a weighted score of 1 to 4. Scores for both the state anxiety and trait anxiety scales can vary from a minimum of 20 to a maximum of 80, where a higher score reflects higher anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Graduate School of Medicine, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided
The datasets generated during and/or analyzed during the current study are not publicly available but are available from the investigators on reasonable request